CLINICAL TRIAL: NCT07077044
Title: Transcutaneous Electrical Nerve Stimulation in Children With Functional Constipation Monitored by Pocket-sized Point-of-care Ultrasound.
Brief Title: The Effects of TTNS, TTNS Combined With PHUS, and Conventional Therapy With PHUS in the Treatment of PFC.
Acronym: constipation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Protocol HMO-0446-23; Hadassah Medical Center trial (Other: Hadassah Medical Center clinical trial)
Record Dates: First submitted 2025-03-17; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-02

CONDITIONS: Constipation; Constipation - Functional
Keywords: children with functional constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: The study will include a convenience sample of 60 children aged 4-14 years who were diagnosed with FC by a physician according to the diagnostic criteria of Rome IV and who had already received treatment for constipation for at least one month, including toilet training and laxative therapy. These will be chosen from the patients visiting the pediatric gastroenterology clinic at Hadassah Medical Center.
  An a priori power analysis (G-Power software, Version 3.1) with the following parameters: 1-β = 0.80, effect size = 0.6, and α = 0.05 was calculated to determine the sample size for comparing the effects of TTNS, TTNS combined with PHUS, and conventional therapy with PHUS. This indicated that a total sample of 48 participants would be needed to detect the main effects. To address the problem of inflated effect size estimates and possible dropout of participants, we will recruit a sample of 60 subjects, 20 subjects for each group. A participant is entitled to withdraw from the study at a
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Arm 1 - TTNS Treatment Only Participants will receive transcutaneous tibial nerve stimulation (TTNS) according to a predefined home-based protocol.
  Arm 2 - TTNS + PHUS Monitoring Participants will receive TTNS as in Arm 1, in combination with periodic monitoring using portable handheld ultrasound (PHUS) to assess rectal parameters.
  Arm 3 - Conventional Treatment + PHUS Monitoring Participants will continue standard pharmacological and behavioral therapy (toilet training and laxatives), monitored by PHUS at regular intervals.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- TTNS treatment with no PHUS assessments (Experimental): TTNS treatment with no PHUS assessments
  Interventions: Device: The transcutaneous posterior tibial nerve stimulation device
- TTNS treatment combined with PHUS assessments (Experimental): TTNS treatment combined with PHUS assessments
  Interventions: Device: The transcutaneous posterior tibial nerve stimulation device; Other: PSUS
- Conventional treatment (Active Comparator): conventional treatment recommendations (medications, diets, and behaviors) previously prescribed by their treating physician.
  Interventions: Other: PSUS

INTERVENTIONS:
Device: The transcutaneous posterior tibial nerve stimulation device — In addition to their conventional treatment, subjects in both TTNS groups will complete eight weeks of home TTNS treatment (3 sessions per week), and each session will last for 20 minutes. Stimulation will be provided by a portable device (Chattanooga®, ContinuumTM, Hixson, TN, USA). The device will be pre-programmed to apply a bi-phasic squared wave with a pulse width of 200μsec, and a pulse frequency of 20 Hz. These are default settings for TTNS that have been used in previous studies for urinary and fecal incontinence59,62,67. Two self-adhesive electrodes (5 x 5 cm) will be placed over the ankle area, one approximately 3 to 4 cm above the medial tibial malleolus and a second electrode just below the medial malleolus of the same leg.
  Arms: TTNS treatment combined with PHUS assessments; TTNS treatment with no PHUS assessments
Other: PSUS — Handheld US
  Arms: Conventional treatment; TTNS treatment combined with PHUS assessments

SUMMARY:
This study is a randomized, controlled trial designed to evaluate the effects of transcutaneous tibial nerve stimulation (TTNS), TTNS combined with pocket-sized handheld ultrasound (PHUS), and conventional therapy with PHUS on children with functional constipation (FC). Participants will be stratified into three intervention arms (n=20 per group).

FC will be defined based on the Rome IV diagnostic criteria, in the absence of organic or anatomical causes. Participants will be between 4 and 14 years old and will have experienced failure of conservative treatment for at least three months prior to enrollment.

The primary outcomes include changes in rectal ultrasound parameters and symptom severity scores. Ultrasound assessments will be conducted by trained clinicians using standardized protocols. Monitoring for adverse events will be performed throughout the intervention phase. Safety considerations include predefined exclusion criteria, such as underlying neurological, metabolic, or cardiac conditions.

DETAILED DESCRIPTION:
Eligibility Criteria

Inclusion Criteria:

Children aged 4 to 14 years.

Diagnosis of functional constipation (FC) established prior to study enrollment. FC is defined according to the Rome IV diagnostic criteria, in the absence of identifiable organic or anatomical causes (e.g., no endocrine, metabolic, anatomical, or neuromuscular dysfunction). No additional diagnostic testing is required for inclusion.

Ability to complete daily diaries and TTNS sessions, either independently or with caregiver support.

Documented failure of conservative medical treatment following at least three months of therapy.

Exclusion Criteria:

Malformations of the digestive system or rectal anatomical anomalies (e.g., large intestinal atresia or stenosis, Hirschsprung's disease, congenital anorectal malformations).

Neurological or psychiatric conditions (e.g., cerebral palsy, spina bifida, intellectual disability, anorexia nervosa).

Major cognitive impairments.

Metabolic disorders (e.g., diabetes mellitus, diabetes insipidus, scurvy, phenylketonuria).

Endocrine disorders (e.g., hypothyroidism).

Cardiovascular conditions such as heart disease or arrhythmias, or presence of ventriculoperitoneal shunts or cardiac pacemakers, due to potential electrical interference.

History of thoracic or abdominal surgery.

Presence of dermatological lesions in the area of electrode application.

Presence of active electronic implants.

ELIGIBILITY:
Inclusion Criteria Children aged 4 to 14 years

Clinical diagnosis of functional constipation (FC), with no identifiable organic or anatomical cause (e.g., endocrine, metabolic, anatomical, or neuromuscular dysfunction)

FC diagnosis established according to Rome IV criteria

No additional tests required to confirm eligibility

Ability to complete daily diaries and TTNS sessions (by participant or caregiver)

Failure of conservative medical treatment (including toilet training and laxatives) after at least three months

Exclusion Criteria Malformations of the digestive system and rectal anatomical anomalies (e.g., large intestinal atresia/stenosis, Hirschsprung's disease, congenital anorectal anomalies)

Neurological or psychiatric disorders (e.g., cerebral palsy, spina bifida, intellectual disability, anorexia nervosa)

Major cognitive impairment

Metabolic conditions (e.g., diabetes mellitus, diabetes insipidus, scurvy, phenylketonuria)

Endocrine disorders (e.g., hypothyroidism)

Cardiac conditions (e.g., heart disease, arrhythmias, presence of pacemaker or ventriculoperitoneal shunt) due to possible interference with electrical stimulation

History of thoracic or abdominal surgery

Presence of skin lesions in the area of electrode application

Presence of active electronic implants

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Severity of constipation using the Wexner Constipation Scoring System (WCSS) | From enrollment to the end of treatment 8 weeks. Then 4 month after this end- will be US final reassessment
  The Wexner Constipation Scoring System (WCSS) will be used to quantify the severity of constipation and evaluate treatment effectiveness. The scale includes 8 items assessing: (1) frequency of defecation, (2) painful defecation, (3) incomplete evacuation, (4) abdominal pain, (5) time per attempt, (6) type of assistance, (7) number of unsuccessful attempts per 24 hours, and (8) duration of symptoms. Items are rated 0-4, except for assistance (0-2), with total scores ranging from 0 to 30 (higher scores = more severe constipation).
  Time Frame:
  Baseline and 4 weeks after intervention start
  Unit of Measure:
  Score on a 0-30 scale
  Secondary Outcome Measures Each outcome must be listed separately, with clear title, description, time frame, and unit.
  1. Stool consistency using the Bristol Stool Form Scale (BSFS) Description: The BSFS classifies stool on a 7-point scale (1 = separate hard lumps; 7 = watery), used to monitor stool consistency.
  Time Frame: Daily entries over 4 weeks Unit of

SECONDARY OUTCOMES:
stool consistency using the Bristol Stool Form Scale (BSFS)77,78 (Appendix 5). The BSFS classifies and categorizes stool consistency on a 7-point scale according to cohesion and surface cracking | 24 hours
  : 1) stool consistency using the Bristol Stool Form Scale (BSFS)77,78 (Appendix 5). The BSFS classifies and categorizes stool consistency on a 7-point scale according to cohesion and surface cracking, as follows: 1, separate hard lumps (like nuts); 2, sausage-shaped but lumpy; 3, like a sausage or snake but with cracks on its surface; 4, like a smooth and soft sausage or snake; 5, soft blobs with a clearcut edge; 6, fluffy pieces with ragged edges and mushy; and 7, watery without solid pieces (1 to 3 indicate constipation; 4-5 is "ideal" stools; 6-7 show paradoxical diarrhea); Numbers of episodes per day will be recorded for 2) defecation; 3) soiling; 4) abdominal pain; 5) presence of bloody stool; A Hebrew version of the visual analog scale (VAS) (Appendix 6) will be used to document a) sensation or urge to defecate79; b) straining and pain during each documented defecation.79 In addition, data on the use of medications for defecation and enemas and/or special diets, as well

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Hebrew University Hospital, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No
: There is currently no plan to share individual participant data (IPD) from this study. The data include sensitive pediatric health information. While de-identification procedures are in place, additional ethical and logistical considerations limit the ability to make IPD publicly available at this stage.

REFERENCES:
- See also: Related Info — https://www.ariel.ac.il/wp/nhpl/